CLINICAL TRIAL: NCT02602483
Title: Randomized, Double Blind, Placebo Controlled Exploratory Study To Assess the Efficacy and Safety of a Triple Combination of Ibuprofen+Mg+Ascorbic Acid for Acute Pain Treatment in Temporomandibular Join Disorder (TMJD) Patients
Brief Title: Exploratory Study To Assess the Efficacy and Safety of a Triple Combination for Acute Pain Treatment in Patients With Temporomandibular Joint Disorders (TMJD).
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spherium Biomed (Industry)
Collaborators: Universitat Internacional de Catalunya (Other); Hospital Odontològic UB (Other); Hospital Universitario La Fe (Other); Hospital Universitario Rey Juan Carlos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JAN12006-01
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-10

CONDITIONS: Temporomandibular Joint Disorders
Keywords: temporomandibular; joint; pain; ibuprofen; magnesium; vitamin C
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain | interventions — Ibuprofen; Magnesium; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Triple combination (Experimental): Powder for oral administration
  Interventions: Drug: Ibuprofen; Drug: Magnesium; Drug: Ascorbic Acid
- Ibuprofen (Active Comparator): Powder for oral administration
  Interventions: Drug: Ibuprofen
- Magnesium + ascorbic acid (Active Comparator): Powder for oral administration
  Interventions: Drug: Magnesium; Drug: Ascorbic Acid
- Placebo (Placebo Comparator): Powder for oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen
  Arms: Ibuprofen; Triple combination
Drug: Magnesium
  Arms: Magnesium + ascorbic acid; Triple combination
Drug: Ascorbic Acid
  Arms: Magnesium + ascorbic acid; Triple combination
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objetive of this study is to explore the efficacy and safety of a triple combination of ibuprofen, magnesium and ascorbic acid for acute pain treatment in TMJD patients

ELIGIBILITY:
Inclusion Criteria:

1. TMD dysfunction syndrome patients of RDC/TMD Groups Ia and/or Ib (+/- IIIa and/or IIIb); with moderate to severe pain (VAS >4), refractory to conservative treatment (including splint / local prosthesis)
2. Subjects between 18 and 65 years.
3. Body weight within the normal range (IMC index between 19 and 30) expressed as weight (kg) /height (m2).
4. Physical condition according to ASA I or II (American Society of Anesthesiologists)
5. Having not participated in previous clinical trial during the three months preceding the setting-up of this study.
6. Free acceptance to collaborate in the study, expressed by signature of written informed consent by the participant

Exclusion Criteria:

1. Patients who are pregnant or breastfeeding.
2. Patients who have a consumption of enzyme-inducing drugs within the 30 days prior to the study: carbamazepinam, nevirapine, phenobarbital, rifampin, secobarbital and St. John's wort.
3. Patients who are consuming: acetaminophen, acetyl salicylic acid, bemiparina, clonixidina, oral anticoagulant, heparin and derivatives, systemic corticosteroids, pemetresed, digoxin, phenytoin, lithium, methotrexate, Salicylates, NSAIDs, antacids containing aluminum, such as algeldrato, magaldrate, morphine and its derivatives.

   Patients who have been medicated with NSAIDs or Morphic derivatives for the treatment of pain of TMD prior to attending the consultation will be included whether, they meet a washout period of 8 to 12 hours (depending on the medication taken) before being included in the study.
4. Patients with underlying systemic pathology candidate to receive drug treatment with analgesic.
5. In patients with a history of gastrointestinal bleeding or perforation related to previous treatment with NSAIDs. Peptic ulcer / active or recurrent gastrointestinal hemorrhage (two or more episodes of ulceration) or proven hemorrhage.
6. Patients with active Ulcerative colitis or Crohn's disease. Severe heart failure. Severe renal dysfunction. Severe hepatic dysfunction.
7. Patients with urolithiasis by oxalate
8. History of alcoholism or drug dependence within 3 months prior to the screening visit, and / or, History of psychotropic drugs consumption within 3 months prior to the screening visit.
9. Heavy consumer of stimulating beverages (>5 coffees, teas, or cola drinks per day).
10. History of drug allergy, idiosyncrasy or hypersensitivity. 11 Patients with cerebrovascular bleeding or other active bleeding 12 Patients with bleeding diathesis or other bleeding disorders .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pain level from baseline compared to placebo assessed by a pain VAS scale | seven days
  Pain level is measured according to visual analogue scale (VAS, 0-100 mm) before and 7 days after treatment.

SECONDARY OUTCOMES:
Change from baseline compared to placebo assessed by RDC/TMD questionnaire at day 3 +/-1 and at day 7. | seven days

CONTACTS AND LOCATIONS:
Overall Officials: Giner Lluis, MD, Principal Investigator — Clinica Universitaria Odontologica de la Universidad Internacional de Cataluña
Locations (4):
- Spain (4):
  - Hospital Odontològic de la Universitat de Barcelona, Barcelona, Barcelona
  - Clinica Universitaria Odontològica de la Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Hospital Universitari i Politècnic La Fe, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided